CLINICAL TRIAL: NCT00396487
Title: Tailored Treatment of Metastatic Colorectal Cancer Based on Genetic Markers
Brief Title: Tailored Treatment in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Only one patient included as per Feb. 4, 2008.
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-2006-002957-56
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; tailored treatment; genetic markers; gene polymorphism; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Irinotecan

INTERVENTIONS:
Drug: Capecitabine, Irinotecan, 5-Fluorouracil+Calciumfolinat

SUMMARY:
To compare the response rate of single agent chemotherapy in advanced colorectal cancer given as standard treatment versus tailored treatment in a randomised phase III trial.

DETAILED DESCRIPTION:
The TS and MTHFR polymorphism has been investigated in a new study based on analysis of normal tissue. The results indicated that protein with a 3/3 TS polymorphism or a MTHFR T polymorphism had a significantly higher response rate and a longer time to progression than the other groups when treated with bolus 5-FU.

Capecitabine is metabolised to 5-FU through a number of enzymatic steps. It is the first rationally designed drug that is based upon the high concentration of thymidine phosphorylase (TP) in many human tumors compared to normal tissue. TP is the last step in the conversion of capecitabine to 5-FU and seems to be the limiting factor for the activation. Capecitabine may to some extent mimic continues 5-FU infusion as opposed to bolus 5-FU. A number of small investigations have indicated that patients with 2R/2R TS polymorphism have a higher response rate than heterozygous patients.

The TS and MTHFR polymorphism analysis can easily be performed on sputum, which means an easy collection and sending of the samples.

At present single agent chemotherapy is based on three drugs (5-FU, capecitabine, and Irinotecan) with almost the same overall activity. It seems rational to investigate if improvement can be obtained by tailoring the treatment according to gene polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* Histopathological verification of the primary tumor
* Measurable disease according to RESIST criteria
* Single agent chemotherapy indicated
* Performance status >=2
* Age >= 60 years
* Life expectancy > 3 months
* Adequate liver and kidney function as evaluated by bilirubin <= 3 times of normal upper limit, ALAT <= 3 times upper normal limit (<= 5 times upper normal limit in case of liver metastases), serum creatinine <= 1.5 times normal upper limit.
* ANC >=1.5 x 109/l and platelets >= 100 x 109/l
* Informed consent

Exclusion Criteria:

* Patients with CNS metastases
* Other malignant disease within the last 5 years except for non-melanoma skin cancer and carcinoma in situ of cervix uteri
* Previous chemotherapy for metastatic disease
* Adjuvant chemotherapy < 6 months before inclusion
* Patients with previous major toxic or allergic reaction to the protocol drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-11; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary end point is
Response according to RECIST criteria.

SECONDARY OUTCOMES:
Secondary end points are
Progression free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, Prof, MDSc, Principal Investigator — Department of Oncology, Vejle Hospital, 7100 Vejle, DK-Denmark
Locations (10):
- Denmark (10):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Hospital Esbjerg, Esbjerg
  - Herlev Hospital, Herlev
  - Herning Central Hospital, Herning
  - Næstved Hospital, Næstved
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Viborg Hospital, Viborg